CLINICAL TRIAL: NCT04964271
Title: Identification and Characterization of Commercial RUO Antibodies for the Detection of Specific Prostate Cancer Tumoral Markers Expressed in Potential Circulating Tumoral Cells (CTCs)
Brief Title: Identification of Prostate Cancer Specific Markers in Patients Compared to Healthy Participants
Status: Active, not recruiting | Type: Observational
Sponsor: Tethis S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: TET-21-002
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer biomarker; circulating tumoral cell; immunofluorescence assay; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low risk prostate cancer patients: Prostate cancer risk category is based on the definition of the European Association of Urology, namely low risk (PSA (prostate-specific antigen) <10 ng/ml, and stage T1/T2a and Gleason score 3+3).
- High risk prostate cancer patients: Prostate cancer risk category is based on the definition of the European Association of Urology, namely high risk (PSA (prostate-specific antigen) >20 ng/ml or stage T3 or higher or biopsy Gleason score 8-10).
- Healthy donor: Participants who are in good health and without history of cancer disease.

SUMMARY:
This is an exploratory research study with the aim of identifying specific cancer biomarkers in various subtypes of prostate cancer. Blood samples will be collected from 60 participants divided into 40 patients and 20 healthy donors.

DETAILED DESCRIPTION:
In this research study different commercial RUO (Research Use Only) antibodies will be purchased and then tested on blood samples obtained by patients affected by prostate cancer and by healthy participants as control. Sixty participants will be enrolled belonging to different risk categories:20 participants affected by prostate cancer at low risk, 20 participants affected by prostate cancer at high risk, and 20 participants without a cancer disease (healthy volunteers) as control.

Risk categorization is based on the definition of the European Association of Urology. After signing the informed consent form, participants will be screened to evaluate if they meet the eligibility criteria. If all the criteria are met, participants will be enrolled into the study and will be asked to provide some demographic and other data. A 13 ml blood sample will be collected by the participants and shipped to Sponsor's laboratories, in order to be processed and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give and sign a written informed consent for participation in the study
* Male, aged 18 years or above
* Diagnosed with prostate cancer at low or high risk
* Candidate to active surveillance (in case of low-risk disease) or treatment with curative intent such as radical prostatectomy or radiation therapy (in case of low risk patients not willing to undergo active surveillance or patients with high risk disease)
* Healthy participants undergoing a visit at the site for reason other than cancer diagnosis (including prostate cancer)

Exclusion Criteria:

* History of other malignancies other than prostate cancer (for healthy participants includes also prostate cancer)
* Undergone surgery or treatment for prostate cancer before enrolment
* Presence of known severe coagulation or haematological disorder
* Absence of written signed informed consent for participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from among the people who visit the urology department
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of commercial Antibodies capable of identify specific Prostate Cancer Biomarkers | day 1 : blood collection day
  Qualitative assessment of Staining Positivity for different Prostate Cancer Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Briganti, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
This is a basic research study without an IPD information sharing plan

REFERENCES:
- [Background] Hench IB, Hench J, Tolnay M. Liquid Biopsy in Clinical Management of Breast, Lung, and Colorectal Cancer. Front Med (Lausanne). 2018 Jan 30;5:9. doi: 10.3389/fmed.2018.00009. eCollection 2018. PMID 29441349
- [Background] Rawal S, Yang YP, Cote R, Agarwal A. Identification and Quantitation of Circulating Tumor Cells. Annu Rev Anal Chem (Palo Alto Calif). 2017 Jun 12;10(1):321-343. doi: 10.1146/annurev-anchem-061516-045405. Epub 2017 Mar 6. PMID 28301753
- [Background] Carbone R, Marangi I, Zanardi A, Giorgetti L, Chierici E, Berlanda G, Podesta A, Fiorentini F, Bongiorno G, Piseri P, Pelicci PG, Milani P. Biocompatibility of cluster-assembled nanostructured TiO2 with primary and cancer cells. Biomaterials. 2006 Jun;27(17):3221-9. doi: 10.1016/j.biomaterials.2006.01.056. Epub 2006 Feb 28. PMID 16504283
- [Background] Zanardi A, Bandiera D, Bertolini F, Corsini CA, Gregato G, Milani P, Barborini E, Carbone R. Miniaturized FISH for screening of onco-hematological malignancies. Biotechniques. 2010 Jul;49(1):497-504. doi: 10.2144/000113445. PMID 20615202
- [Background] Krol I, Schwab FD, Carbone R, Ritter M, Picocci S, De Marni ML, Stepien G, Franchi GM, Zanardi A, Rissoglio MD, Covelli A, Guidi G, Scarinci D, Castro-Giner F, Mazzarella L, Doglioni C, Borghi F, Milani P, Kurzeder C, Weber WP, Aceto N. Detection of clustered circulating tumour cells in early breast cancer. Br J Cancer. 2021 Jul;125(1):23-27. doi: 10.1038/s41416-021-01327-8. Epub 2021 Mar 24. PMID 33762721
- [Background] Scher HI, Graf RP, Schreiber NA, McLaughlin B, Jendrisak A, Wang Y, Lee J, Greene S, Krupa R, Lu D, Bamford P, Louw JE, Dugan L, Vargas HA, Fleisher M, Landers M, Heller G, Dittamore R. Phenotypic Heterogeneity of Circulating Tumor Cells Informs Clinical Decisions between AR Signaling Inhibitors and Taxanes in Metastatic Prostate Cancer. Cancer Res. 2017 Oct 15;77(20):5687-5698. doi: 10.1158/0008-5472.CAN-17-1353. Epub 2017 Aug 17. PMID 28819021
- [Background] Xu L, Jia S, Li H, Yu Y, Liu G, Wu Y, Liu X, Liu C, Zhou Y, Zhang Z, Sheng Y. Characterization of circulating tumor cells in newly diagnosed breast cancer. Oncol Lett. 2018 Feb;15(2):2522-2528. doi: 10.3892/ol.2017.7540. Epub 2017 Dec 6. PMID 29434968
- [Background] Roviello G, Corona SP, Bonetta A, Cappelletti MR, Generali D. Circulating tumor cells correlate with patterns of recurrence in patients with hormone-sensitive prostate cancer. Onco Targets Ther. 2017 Jul 31;10:3811-3815. doi: 10.2147/OTT.S143020. eCollection 2017. PMID 28814879